CLINICAL TRIAL: NCT05437705
Title: Decoding and Modulating Affective Brain States
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Desmond Oathes, Assistant Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 850664
Record Dates: First submitted 2022-06-13; First posted 2022-06-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Rumination; Major Depressive Disorder; Anxiety
Keywords: TMS; rumination; depression; anxiety
MeSH Terms: conditions — Rumination Syndrome; Depressive Disorder, Major; Anxiety Disorders; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All subjects will receive TMS using the optimized and least optimized frequencies, but the order is randomized and counterbalanced.
Who Masked: Participant
Masking Description: The study will use a single-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Neuromodulation using the optimal rTMS stimulation frequency (Experimental): Through manipulation of brain state with a negative-affect task and using fMRI as the feedback signal, the investigators aim to fine-tune repetitive Transcranial Magnetic Stimulation (rTMS) delivery to maximally impact the desired brain states in awake, behaving participants in a highly individualized manner (Visit 3). The optimal rTMS stimulation frequency will then be tested in a 3-day rTMS neuromodulation intervention.
  Interventions: Device: Transcranial Magnetic Stimulation
- Neuromodulation using the least optimal rTMS stimulation frequency (Active Comparator): The investigators will compare the results of the optimal rTMS frequency neuromodulation with a separate 3-day neuromodulation session using the least optimal rTMS frequency, as determined by the results of Visit 3.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication. The MagPro X100* magnetic stimulator and Cool-B65 Butterfly Coil are FDA-approved for rTMS treatments of depression.

SUMMARY:
The research study is being conducted to study brain patterns of negative emotion and develop personalized brain stimulation protocols to disrupt these patterns with transcranial magnetic stimulation (TMS). First, the investigators will use functional Magnetic Resonance Imaging (fMRI) data to generate a negative affect map for each participant. Then, the investigators will apply a variety of repetitive transcranial magnetic stimulation (rTMS) sequences while the participant is inside the MRI scanner to determine the optimal and least optimal rTMS frequencies at changing negative affect brain states. Finally, these two frequencies will be tested over two 3-day rTMS neuromodulation sessions to assess whether they can reduce negative emotions.

DETAILED DESCRIPTION:
The study involves 11 visits over approximately 10 weeks, depending on scanner availability and scheduling. See below for the study schedule with a summary of the procedures:

* Visit 1: Screening Procedures (~3-4 hours). The first part of the screening will take place remotely (~1 hour). The investigators will begin by reviewing the Informed Consent Form (ICF). Participants who agree to participate and sign the ICF will then complete several questionnaires. Those who meet preliminary eligibility criteria based on the remote procedures will be invited for an in-person visit. The in-person screening will include a brief TMS demonstration (~20 minutes). If TMS is well tolerated, the visit will proceed to a comprehensive clinical interview (~2-3 hours) to assess current and past mental health history.
* Visit 2: Baseline MRI & Assessments (~2 hours). This visit will involve a 1-hour MRI scan, including both structural and functional sequences, and an assessment session with computerized tasks and questionnaires.
* Visit 3: MRI Scan with TMS (~2.5 hours). A second MRI scan will be conducted with concurrent TMS procedures. Participants will complete a mental task while interleaved rTMS is delivered at different frequencies. This scan will be used to determine the optimal stimulation frequency for each participant.
* Visits 4-6: First Neuromodulation Session (~1.5 hours each). Participants will receive rTMS using either the optimal or least optimal stimulation frequency. They will also complete two computerized tasks after rTMS, with questionnaires in between procedures.
* Visit 7: MRI Scan with TMS (~2 hours). This visit will be a shortened version of Visit 3, as some MRI scans and questionnaires will not need to be repeated.
* Visits 8-10: Second Neuromodulation Session (~1.5 hours each). These visits will mirror Visits 4-6. However, the TMS condition administered (optimal or suboptimal frequency) will be counterbalanced with the condition used during the first neuromodulation session. Visit 8 will be scheduled at least 2 weeks after Visit 7.
* Visit 11: MRI Scan with TMS (~2 hours). This visit will mirror Visit 7.

After completing all procedures, participants will receive the full study compensation. Payments may be issued earlier if participants request compensation after each visit or if they withdraw early.

ELIGIBILITY:
Inclusion criteria:

1. 18-65 years old
2. Patient Health Questionnaire (PHQ-9 score) = or > than 10
3. Comprehension of instructions in the English language.
4. Capacity to provide informed consent and follow study procedures.
5. Availability for the duration of the study.

Exclusion Criteria:

1. Diagnosis of bipolar disorder (as PI discretion), schizophrenia or other psychotic disorder
2. Recent use of psychoactive medications or substances as determined by investigators
3. History of neurological disorder or traumatic brain injury (other than mild)
4. Unable to have an MRI scan, or current or prior medical condition that could interfere with the collection or interpretation of MRI data
5. Unable to receive or tolerate TMS
6. Implanted devices, such as an aneurysm clip or cardiac pacemaker
7. History of stroke, epilepsy, or brain scarring
8. Pregnant, nursing, or trying to become pregnant (self-attestation alone)

During this study, participants are asked to:

1. Refrain from substance use (including marijuana and illicit drugs) for duration of the study (self-attestation alone).
2. Abstain from alcohol for 24 hours before the MRI scans (self-attestation alone).
3. Abstain from increasing caffeine intake or begin taking any new medications (self-attestation alone).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in ruminative response scale (RRS) score after using the optimal rTMS stimulation frequency vs the least optimal rTMS stimulation frequency | Up to 4 weeks
  By comparing the RRS score change pre/post rTMS of both neuromodulation sessions (Visits 4-6/7-9) the investigators will determine whether the optimal rTMS stimulation frequency is more effective at improving clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Oathes, PhD, Principal Investigator — Associate Professor of Psychiatry
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States